CLINICAL TRIAL: NCT07155239
Title: 1726-nm Laser (AviClear) for Hidradenitis Suppurativa (HS): A Randomized Split-Body, Sham-Controlled Pilot Trial
Brief Title: 1726-nm Laser for Acne Inversa (Hidradenitis Suppurativa)
Acronym: WMCREI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wynn Medical Center (Other)
Responsible Party: Principal Investigator, Huynh Wynn Tran MD FACP, CEO/Founder, Wynn Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: WMCREILAS082025
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: hidradenitis suppurative; inversa acne
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Arm (Sham Comparator): handpiece contact, no cooling, no energy
  Interventions: Device: Sham (No Treatment)
- Laser Treatment (Experimental): Laser treatment three sessions at Weeks 0, 4, 8; follow-ups at Weeks 12, 16, 24.
  Interventions: Device: AviClear Lase Treatment

INTERVENTIONS:
Device: AviClear Lase Treatment — Three laser sessions at Weeks 0, 4, 8; follow-ups at Weeks 12, 16, 24.
  Arms: Laser Treatment
Device: Sham (No Treatment) — No active laser treatment
  Arms: Control Arm

SUMMARY:
Hidradenitis suppurativa (HS) is a long-lasting skin condition that causes painful lumps, abscesses, and tunnels in areas such as the armpits and groin. HS begins around the hair follicle; when the follicle becomes blocked and inflamed, new lesions form. Prior clinical studies of lasers that act on the hair follicle have shown improvement in HS symptoms, and a 1726-nm diode laser-designed to selectively heat oil glands within the follicle-has reduced inflammatory lesions in acne with good tolerability across many skin types.

This study will test whether a 1726-nm diode laser can safely reduce inflammatory HS lesions in Hurley stage I-II disease. Adults with bilateral (right/left) affected areas will be randomized so that one side receives active laser treatment and the other side receives a sham procedure. Participants will have three treatment sessions over 8 weeks and follow-up through Week 24 while continuing their stable HS medications.

The primary outcome is the percent change in abscess and inflammatory nodule counts on the treated side versus the sham side at Week 16. Secondary outcomes include validated HS responder scores, pain, quality of life, flare rate/antibiotic use, and safety. Results may support a non-ablative, follicle-directed option for early HS.

DETAILED DESCRIPTION:
Hidradenitis suppurativa (HS) is a chronic, relapsing inflammatory disorder of the hair follicle characterized by painful nodules, abscesses, and dermal tunnels that cluster in intertriginous sites. Contemporary models place follicular occlusion and rupture of the pilosebaceous unit, rather than primary apocrine disease, at the start of the cascade, with downstream innate/adaptive immune activation (e.g., TNF-α, IL-17/IL-23 axes). This follicle-centric pathogenesis underpins the therapeutic logic for energy-based approaches that target follicular structures to reduce lesion initiation.

Multiple controlled studies show that laser/light devices aimed at the folliculo-sebaceous apparatus can improve HS activity, supporting this mechanistic rationale. In a randomized controlled trial (n=22) of long-pulsed 1064-nm Nd:YAG, three monthly sessions reduced HS severity (modified HS-LASI) by ~65% overall at 3 months in treated vs control sites (p<0.02), with site-specific reductions (inguinal ~73%, axillary ~62%).

As the investigators noted, the success of a hair-epilation laser reinforces primary follicular involvement in HS. Beyond Nd:YAG, laser hair-removal (LHR) platforms have also demonstrated efficacy. A randomized controlled trial of 755-nm alexandrite LHR in mild-to-moderate HS showed improvements on validated clinical measures (e.g., HiSCR), with acceptable safety, again pointing to the clinical relevance of follicular targeting in reducing inflammatory lesion burden and flares.

Parallel evidence from acne, another follicular occlusion disease, motivates us to investigate 1726-nm (AviClear) sebaceous-selective photothermolysis for HS. Preclinical modeling and in-vivo histology demonstrate that 1726 nm + contact cooling can deliver selective thermal injury to sebaceous glands while sparing surrounding tissue, achieving the canonical endpoint of selective photothermolysis. Clinically, 1726-nm laser studies in acne report significant reductions in inflammatory lesion counts after a short series of treatments, durable improvement at longer follow-up, and favorable tolerability across Fitzpatrick I-VI.

Translating this to HS is biologically plausible for Hurley I-II disease, where new nodule formation remains dominated by follicular events rather than extensive sinus tracts. By reducing sebaceous output and follicular activity, 1726-nm treatment may decrease the frequency and intensity of inflammatory nodules/abscesses, complementing stable background medical therapy (e.g., antibiotics, hormones, or biologics targeting TNF-α/IL-17). Importantly, while energy-based surgery (e.g., CO₂ laser deroofing) is effective for chronic tunnels, a non-ablative, follicle-directed device could address earlier lesional biology, potentially lowering flare rates and delaying progression to scarring disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-60 years; any sex; Fitzpatrick I-VI.
* Clinical HS, Hurley I-II (Investigator confirmed).
* At least one inflammatory nodule in a paired, bilateral region (axilla, groin/inguinal, inframammary, inner thigh, or buttock) within 4 weeks prior to baseline.
* Able to read/speak English/Chinese/Spanish/Vietnamese and sign consent.
* Willing/able to comply with visits, pre/post-care, standardized photography.
* Agree to avoid new HS procedures/therapies in study areas through Week 24.
* No laser contraindication; agrees to shave/clip hair before treatments.
* Optional translational cohort: willing to undergo 4-mm punch biopsy at baseline and Week 16 from the randomized regions (separate consent).

Exclusion Criteria:

* Hurley III (extensive sinus tracts).
* No qualifying nodule(s) in paired bilateral regions in past 4 weeks.
* Prior device/procedure to target areas within 3 months (chemical peel, dermabrasion, microneedling/RF, other lasers/LBB, cryo/chemo-destruction)
* Had Botulinum toxin in target areas within 3 months or planned during study.
* Had systemic retinoid (e.g., isotretinoin) within 3 months.
* Photosensitizing meds that, in PI's judgment, materially increase risk and cannot be held.
* Pregnancy/breastfeeding/plans to conceive during study.
* Active infection, still healing wounds (investigator judgment) in target areas.
* History of keloids/hypertrophic scars, radiation to target areas, malignancy in target areas, diagnosed immunodeficiency, uncontrolled coagulation disorder or therapeutic anticoagulation that cannot be safely managed.
* Excessive tanning or inability to avoid tanning.
* Any condition (medical/mental) or prisoner status that in PI's opinion compromises safety or adherence.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent change from HS baseline | 16 weeks
  Percent change in abscess and inflammatory nodule (AN) count from baseline on the treated side versus the sham side (split-body comparison). HiSCR25 is defined as ≥25% reduction in AN count from baseline, with no increase in abscesses or draining fistulas.
Change in pain | 16 weeks
  Change in pain as measured by the Visual Analogue Scale (VAS), ranging from 0 to 10, with higher scores indicating greater pain

SECONDARY OUTCOMES:
Change in depression scale | 16 weeks
  Change in depression as measured by the Patient Health Questionnaire-9 (PHQ-9), a validated nine-item instrument that assesses depression severity over the preceding 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Huynh Wynn Tran CEO/Founder, MD FACP, Principal Investigator — Wynn Medical Center Research and Education Institute; Molynna Nguyen Clinical Research Manager, BS, Study Director — Wynn Medical Center Research and Education Institute
Locations (1):
- Wynn Medical Center Rheumatology/Dermatology, Rosemead, California, United States

IPD SHARING:
Plan to Share IPD: Yes
demographic and general information
Supporting Information: Study Protocol, SAP
Time Frame: 08/2025 to 12/2026
Access Criteria: similar studies and prior approval from our institution